CLINICAL TRIAL: NCT06365086
Title: Targeting Personalized Brain States Reflecting Strong and Weak Corticospinal Tract Output in Real-time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00000608
Record Dates: First submitted 2024-04-05; First posted 2024-04-15 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Neurotypical Adults

STUDY DESIGN:
Intervention Model Description: Participants will receive single-pulse TMS during personalized brain activity patterns reflecting either strong or weak corticospinal tract activation
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Personalized brain state-dependent single-pulse TMS — Single-pulse TMS will be applied to the right hemisphere during brain activity patterns associated with strong and weak corticospinal tract activation. Single-pulse TMS will also be applied to the right hemisphere during random brain activity patterns.

SUMMARY:
Transcranial magnetic stimulation (TMS) interventions could feasibly strengthen residual corticospinal tract (CST) connections and enhance recovery of paretic hand function after stroke. To maximize the therapeutic effects of such interventions, they must be delivered during poststroke brain activity patterns during which TMS best activates the residual corticospinal tract and enhances neural transmission within it (i.e., brain state-dependent TMS). In this study, the investigators will test the feasibility of real-time, personalized brain state-dependent TMS in neurotypical adults.

Participants will visit the laboratory for one day of testing. Upon arrival, participants will provide their informed consent; afterwards, they will complete eligibility screening. The investigators will then place recording electrodes on the scalp using a swim-type cap and on the left first dorsal interosseous, abductor pollicis brevis, and extensor digitorum communis muscles. After determining the location at which TMS best elicits muscle twitches in the left first dorsal interosseous, the investigators will determine the lowest possible intensity at which TMS elicits muscle twitches at least half of the time in this muscle. Then, the investigators will deliver 6 blocks of 100 single TMS pulses while the participant rests quietly with their eyes open; stimulation will be delivered at an intensity that is 20% greater than the lowest possible intensity at which TMS elicits muscle twitches at least half of the time. Afterwards, the investigators will use the muscle and brain activity recordings acquired during these 6 blocks to build a personalized mathematical model that identifies which patterns of brain activity correspond to the largest TMS-evoked muscle twitches. The investigators will then use this model to detect the occurrence of these brain activity patterns in real-time; when these patterns are detected, single TMS pulses will be delivered. Afterwards, all recording electrodes will be removed, participation will be complete, and participants will leave the laboratory.

The investigators will recruit a total of 16 neurotypical adults for this study.

ELIGIBILITY:
Inclusion Criteria:

* Right-hand dominance
* Willingness to participate
* Ability to provide informed consent

Exclusion Criteria:

* History of major neurological, orthopedic, psychiatric, or cardiovascular disease
* Presence of contraindications to transcranial magnetic stimulation (TMS) or peripheral nerve stimulation (PNS), including:

  * history of adverse reactions to TMS or PNS
  * history of stroke or head injury
  * metal in head, eyes, neck, chest/trunk, or arms, including but not limited to shrapnel,
  * surgical clips, fragments from metalworking, fragments from welding
  * implanted devices
  * history of frequent and severe headaches or migraines
  * immediate family history of seizure or epilepsy
  * personal history of seizure or epilepsy
  * current, suspected, or planned pregnancy
  * current or recent (within the last 3 months) use of medications acting on the central nervous system, including but not limited to: antipsychotic drugs, antidepressants, benzodiazepines, prescription stimulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Result] Khatri UU, Pulliam K, Manesiya M, Cortez MV, Millan JDR, Hussain SJ. Personalized whole-brain activity patterns predict human corticospinal tract activation in real-time. Brain Stimul. 2025 Jan-Feb;18(1):64-76. doi: 10.1016/j.brs.2024.12.1193. Epub 2024 Dec 21. PMID 39716573
- See also: Raw data — https://openneuro.org/datasets/ds005779/versions/1.0.1
- See also: Analysis code — https://github.com/SMNPLab/Realtime_decoding_neurotypical.git

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no specific pre-assignment procedures or events for this study.
Groups:
- Healthy Adults: Healthy adults first had single-pulse TMS delivered to the right motor cortex irrespective of ongoing brain activity (i.e., brain states) in order to generate a training dataset that included brain activity recordings and muscle responses to TMS delivery.
  Then, this training dataset was used to build a personalized mathematical model that discriminated between brain activity patterns reflecting strong and weak corticospinal tract (CST) activation (i.e., strong and weak CST states).
  After building this model, participants received single-pulse TMS to the right motor cortex during personalized brain states reflecting strong corticospinal tract (CST) activation (strong CST states), weak CST states, and random CST states. Stimulation was delivered at 120% of resting motor threshold and motor-evoked potentials (MEPs) were recorded from the left first dorsal interosseous muscle.
Period: Training Phase
Arm/Group | Healthy Adults
Started | 21
Completed | 21
Not Completed | 0
Period: Testing Phase
Arm/Group | Healthy Adults
Started | 21
Strong CST States | 21
Weak CST States | 21
Random CST States | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Adults: Healthy adults received single-pulse TMS the right motor cortex during personalized brain states reflecting strong corticospinal tract (CST) activation (strong CST states), weak CST states, and random CST states. Stimulation was delivered at 120% of resting motor threshold and motor-evoked potentials (MEPs) were recorded from the left first dorsal interosseous muscle.
Arm/Group | Healthy Adults
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (3.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 3
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Motor-evoked Potential (MEP) Amplitudes
Description: Peak-to-peak MEP amplitudes elicited by single transcranial magnetic stimulation (TMS) pulses delivered during personalized strong and weak CST states will be measured from the left first dorsal interosseous muscle. At the individual participant level, all MEP amplitudes will be normalized to the mean MEP amplitude observed in that participant. Mean normalized MEP amplitudes will be compared across CST states.
Time Frame: single session
Measure: Mean (Standard Error); unit: arbitrary units (normalized microvolts)
Groups:
- Strong CST States: Normalized MEPs elicited during strong CST states were calculated.
- Weak CST States: Normalized MEPs elicited during weak CST states were calculated.
- Random CST States: Normalized MEPs elicited during random CST states were calculated.
Arm/Group | Strong CST States | Weak CST States | Random CST States
Number analyzed (Participants) | 19 | 19 | 19
arbitrary units (normalized microvolts) | 1.13 (0.05) | 0.96 (0.04) | 0.90 (0.05)

2. Secondary Outcome: State-targeting Accuracy
Description: An offline version of the real-time EEG analysis algorithm will be used to determine the brain state (i.e., strong or weak CST states, or neither) immediately preceding delivery of each single TMS pulse. The proportion of trials during which the online and offline versions of the real-time EEG analysis algorithm produce the same brain state prediction will be calculated per participant and used as a state-targeting accuracy metric. State-targeting accuracy metrics will be compared to the theoretical chance level (0.5).
Time Frame: single session
Measure: Mean (Standard Error); unit: percentage of trials accurately targeted
Groups:
- Strong CST States: The ability of our real-time system to accurately target strong CST states was calculated.
- Weak CST States: The ability of our real-time system to accurately target weak CST states was calculated.
- Random CST States: Due to the nature of this condition, the ability of our real-time system to accurately target random CST states cannot be calculated.
Arm/Group | Strong CST States | Weak CST States | Random CST States
Number analyzed (Participants) | 19 | 19 | 19
percentage of trials accurately targeted | 94.5 (1.1) | 89.5 (2.7) | NA (NA) — Due to the nature of this condition, the ability of our real-time system to accurately target random CST states cannot be calculated.

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 day
Arm/Group | Healthy Adults
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT06365086/Prot_SAP_003.pdf
  • Informed Consent Form (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT06365086/ICF_002.pdf